CLINICAL TRIAL: NCT05230316
Title: Recognizing Gynecological Symptoms and Health-related Quality of Life in Egyptian Women With Systemic Lupus Erythematosus
Brief Title: Gynecological Symptoms and Health-related Quality of Life in Egyptian Women With SLE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, rehab abdelhamid aboshama, lecturer of obstetrics and gynecology Faculty of medicine, Fayoum University
Other Study IDs: R 205
Record Dates: First submitted 2022-01-05; First posted 2022-02-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: SLE; Menstrual Irregularity
Keywords: SLE; Menstrual irregularity; quality of life
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of our study was to Recognize gynecological symptoms and health-related quality of life in Egyptian women with systemic lupus erythematosus and evaluate the impact of duration of remission on QOL in SLE patients.

DETAILED DESCRIPTION:
Despite significant advances in recent decades, systemic lupus erythematosus (SLE) is still burdened by irreversible organ damage and a notable impact on health-related quality of life (HRQoL). Improving the quality of life is a pivotal goal in the management of SLE. According to the Treat to Target (T2T) recommendations for SLE management, particular attention needs to be paid to the factors that negatively influence HRQoL such as fatigue, pain and depression.

Recent epidemiological studies demonstrate that prolonged remission is an achievable target in SLE patients and is clearly associated with better outcomes in terms of damage accrual. Such findings also raise questions about the possible impact of remission on HRQoL. In a retrospective study, Patients in prolonged remission reported significantly better HRQoL as assessed by the 36-Item Short-Form Health Survey (SF36) and Lupus PRO questionnaire.

Methodology in details L:

70 women with SLE will be included in this study from the outpatient clinic. in Fayoum University hospital It will be conducted in the Department of Obstetrics and Gynecology, Fayoum University Maternity Hospital, Egypt.

Full history taking (Age, Duration of marriage, Parity, Occupation, Mode of delivery, History of abortion, Medical and Surgical history).

Menstrual histories obtained from participants included: age at menarche, duration of heavy bleeding, duration of menses and menstrual cycle, and other gynecological symptoms as Questionnaire form.

Patients' blood pressure, height, weight, body mass index (BMI), and other clinical parameters were reviewed by the attending doctors.

The patient's medications, which included immunosuppressive therapy such as steroids, cyclophosphamide, azathioprine, and cyclosporine A, where noted, and the use of other adjunctive medications were also recorded.

Definition of remission Definition of remission was in line with European Consensus Criteria . Clinical remission (CLR) was present when clinical SLEDAI score=0 and physician global score less than 0.5

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilling the American College of Rheumatology (ACR) 1982 revised criteria for SLE,
2. age between 15 and 55 years
3. and consented to the interview.

Exclusion Criteria:

1. Patients with active malignancy
2. and end-stage lupus nephritis
3. Patients who had been treated with Belimumab in the last 7 years, due to the reported effects of Belimumab on HRQoL.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 70 women with SLE will be included in this study from the outpatient clinic. in Fayoum University hospital It will be conducted in the Department of Obstetrics and Gynecology, Fayoum University Maternity Hospital, Egypt, and department of rheumatology Assiut university Assiut Egypt
  The study protocol was approved by the medical research and ethics committee of the institution, and written informed consent was obtained from all subjects. Patients fulfilling the American College of Rheumatology (ACR) 1982 revised criteria for SLE, aged between 15 and 55 completed years, were enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Recognize gynecological symptoms in Egyptian women with systemic lupus erythematosus. | 3 month
  Normal menstrual pattern duration of each menses was between five and 13 days, and the menstrual cycle was between 21 and 35 days. Menarche was defined as the first menstrual period. Oligomenorrhoea was defined as menses occuring at intervals longer than 35 days. Secondary amenorrhoea was defined as the cessation of menses after menstrual cycle has begun and lasted for at least four months for patients with regular cycles, or for at least three of the previous three cycle intervals for patients with irregular cycles.(4) Transient amenorrhoea was defined as when patients resumed her own "normal" cycle after episodes of amenorrhoea, and sustained amenorrhoea was when the patient remained amenorrhoeic until the interview date.
Recognize health related quality of life in Egyptian women with systemic lupus erythematosus. | 3 months
  According to the Treat to Target (T2T) recommendations for SLE management, particular attention needs to be paid to the factors that negatively influence HRQoL such as fatigue, pain and depression.

SECONDARY OUTCOMES:
Evaluate the impact of duration of remission on QOL in SLE patients. | 3 months
  Clinical remission (CLR) is present when clinical SLEDAI score=0

CONTACTS AND LOCATIONS:
Overall Officials: Laila E Abdelfattah, Ass. prof, Study Director — Associated professor of obestatrics and gynecology Faculty of medicine Fayoume university; rehab A aboshama, lecturer, Principal Investigator — lecturer of obstetrics and gynecology
Locations (2):
- Egypt (2):
  - Fayoum university faculity of medicine, Al Fayyum, Fayoum University Zone
  - Fayoum university, Al Fayyum

IPD SHARING:
Plan to Share IPD: No